CLINICAL TRIAL: NCT06125743
Title: Promoting Self-Management in Head and Neck Cancer Survivors With Lymphedema and Fibrosis [PROMISE Trial]
Brief Title: Self-Management for Head and Neck Lymphedema and Fibrosis [PROMISE Trial]
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC# 12323
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema of the Head and Neck
Keywords: Lymphedema; Fibrosis; Head and Neck Cancer; Survivorship; Self-Management
MeSH Terms: conditions — Lymphedema; Fibrosis; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Other)
  Interventions: Behavioral: Usual Care
- In-Person LEF-SMP (Experimental)
  Interventions: Behavioral: In-Person LEF-SMP
- Telehealth LEF-SMP (Experimental)
  Interventions: Behavioral: Telehealth LEF-SMP

INTERVENTIONS:
Behavioral: Usual Care — Participants will conduct self-care activities prescribed by their treating lymphedema therapists.
  Arms: Usual Care
Behavioral: In-Person LEF-SMP — Participants will receive the in-person LEF-SMP intervention.
  Arms: In-Person LEF-SMP
Behavioral: Telehealth LEF-SMP — Participants will receive the telehealth LEF-SMP intervention.
  Arms: Telehealth LEF-SMP

SUMMARY:
The goal of this study is to evaluate the effectiveness of a standardized lymphedema and fibrosis self-management program (LEF-SMP) to improve LEF self-management and reduce LEF-associated symptom burden, functional deficits, and improve quality of life in head and neck cancer (HNC) survivors.

DETAILED DESCRIPTION:
In HNC survivors with lymphedema and fibrosis (LEF), the investigators will: 1) compare the effects of in-person LEF-SMP, telehealth LEF-SMP, and usual care on LEF severity; 2) compare the effects of in-person LEF-SMP, telehealth LEF-SMP, and usual care on LEF-related symptom burden, functional impairments, and quality of life; and 3) compare the effects of in-person LEF-SMP, telehealth LEF-SMP, and usual care on LEF-related knowledge, skills, self-efficacy, and self-care adherence.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Post HNC primary treatment
* No evidence of cancer (NED)
* Completion of initial lymphedema therapy for head and neck lymphedema
* Unable to obtain lymphedema therapy due to barriers noted above
* History of lymphedema on the face and neck, with or without fibrosis
* Ability to understand English in order to complete questionnaires
* Ability to perform self-care activities for LEF management
* Ability to provide informed consent
* Having an electronic device (a computer, tablet, iPad, or smartphone) and internet access at home
* A valid email address

Exclusion Criteria:

* Recurrent or metastatic cancer
* Any other active cancer
* Acute infection
* Acute congestive heart failure
* Acute renal failure
* Cardiac or pulmonary edema
* Sensitive carotid sinus
* Severe carotid blockage
* Uncontrolled hypertension
* Venous thrombosis
* Pregnant people
* Incarcerated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in severity of lymphedema and fibrosis | Baseline, 3-, 6-, and 9-months post-intervention
  This outcome measure will be assessed via Head and Neck - External Lymphedema and Fibrosis Assessment Criteria (HN-LEF Assessment Criteria). The total severity score of lymphedema and fibrosis (LEF) is calculated by summing the severity score (normal = 0, mild =1, moderate =2, and severe =3) of each anatomical site affected by head and neck LEF. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in severity of symptom burden | Baseline, 3-, 6-, and 9-months post-intervention
  This outcome measure will be assessed via Head and Neck - Lymphedema and Fibrosis Symptom Inventory (HN-LEF Symptom Inventory). The severity score of symptom burden is dependent on the number of self-reported symptoms [overall score range: 0 (no) - 5 (severe)], and higher scores mean a worse outcome.
Changes in degrees of jaw range of motion | Baseline, 3-, 6-, and 9-months post-intervention
  This outcome measure will be assessed via Jaw Range of Motion Scale. Higher degrees of jaw range of motion mean a better outcome (criteria for trismus: mouth opening < 35mm).
Changes in degrees of cervical range of motion | Baseline, 3-, 6-, and 9-months post-intervention
  This outcome measure will be assessed via Cervical Range of Motion Instrument. Higher degrees of cervical range of motion mean a better outcome.
Changes in quality-of-life score | Baseline, 3-, 6-, and 9-months post-intervention
  This outcome measure will be assessed via European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This questionnaire includes a global health-related quality of life scale, 5 functional subscales, 3 symptom scales, and 6 single items. Scores for all scales and single items are linearly converted to range from 0-100, and higher scores signify a higher quality of life.
Changes in LEF-related knowledge score | Baseline, 3-, 6-, and 9-months post-intervention
  LEF-related knowledge will be assessed via HN-LEF Knowledge Test scale. The scale asks participants to answer 35 true/false questions. The total score (score range: 0-35) represents participants' knowledge level related to head and neck LEF, and higher scores mean a better outcome.
Changes in LEF-related skills | Baseline, 3-, 6-, and 9-months post-intervention
  LEF-related skills will be assessed via HN-LEF Skill Checklist. Study lymphedema therapists use this checklist to evaluate participants' LEF self-care skills.
LEF-related self-efficacy score | Baseline, 3-, 6-, and 9-months post-intervention
  LEF-related self-efficacy will be assessed via Perceived Medical Condition Self-Management Scale [8-item, each item score 1 (strongly disagree) - 5 (strongly agree)]. Higher scores indicate greater self-efficacy.
LEF-related self-care adherence status | Baseline, 3-, 6-, and 9-months post-intervention
  LEF-related self-care adherence will be assessed via LEF Self-Care Checklist. Higher scores indicate greater better adherence to LEF self-care activities (i.e., full adherence: ≥ 5 days; partial adherence: 3-4 days; non-adherence: <3 days).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Barbara Murphy, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng J, Abene J, Huang L, Murphy BA. Study protocol for a multi-site randomized clinical trial of an intervention program to promote self-management among head and neck cancer survivors with lymphedema and fibrosis [PROMISE trial]. Trials. 2025 Oct 13;26(1):404. doi: 10.1186/s13063-025-09089-x. PMID 41084063